CLINICAL TRIAL: NCT02101762
Title: A Clinical Study to Compare the CAUTI Rates Following ERASE CAUTI Tray Non-Silver Coated Foley Catheters Verse Silver Coated Foley Catheters
Brief Title: Study to Compare CAUTI Rates Following ERASE CAUTI Tray Non-Silver vs Silver Coated Foley Catheters
Status: Terminated | Type: Observational
Why Stopped: Funding
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Other Study IDs: MII-001
Record Dates: First submitted 2012-02-09; First posted 2014-04-02 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Surgery; Intensive Care Units
Keywords: Foley; Catheters; CAUTI; ERASE CAUTI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Silver Coated Catheters: Subjects that had previously received silver coated Foley catheters.
- ERASE CAUTI Non-Silver Coated Catheters: Subjects that received non-silver catheters from an ERASE CAUTI tray.

SUMMARY:
The Foley catheter is one component in a catheter insertion procedure that could contribute to a catheter associated urinary tract infection (CAUTI). Improvement in the catheter insertion procedures using the ERASE CAUTI Tray system may help to lower these infection rates.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Received Either silver coated Foley catheter or ERASE CAUTI non-silver coated catheter

Exclusion Criteria:

* UTI present upon current hospital admission
* Burn patients, transplant patients, or immune-compromised patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring urinary Foley catheters.
Sampling Method: Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Urinary tract infection rates | 3-9 months based on size of ICU and catheter usage
  Infection rate/1000 catheter days.

SECONDARY OUTCOMES:
Catheter use | Catheter days
  Number of days catheters used.
Infection Costs | Duration of infection
  Catheter related charges for infections

CONTACTS AND LOCATIONS:
Overall Officials: Ed Drower, MS, Study Director — Medline Industries

IPD SHARING:
Plan to Share IPD: No